CLINICAL TRIAL: NCT05044559
Title: Effect of Continuous Positive Airway Pressure in Phase 1 Cardiac Rehabilitation After Post CABG
Brief Title: Continuous Positive Air Way Pressure in Cardiac Rehabilitation After CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00593 Memoona Salal
Record Dates: First submitted 2021-09-13; First posted 2021-09-14 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Post-cardiac Surgery
Keywords: Continuous Positive Airway Pressure; Coronary Artery Bypass Graft Surgery; Inpatients Rehabilitations
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Positive Air Way Group (Experimental): Day 1: Use of CPAP between 10 and 12 cmH2O according to tolerance for 20 minutes two time a day at first day of post surgery bed mobility chest physiotherapy ,active assistive ROM 5 repetitions of upper and lower limb, ACBT cycle. ABGS was analyses at first minute of exercise. and vital was record after exercise.
  Day 2: Active ROM exercise progress of 5 repetitions bed to chair mobility. same exercise progress with 5 repetition and 5 minute walk( day 3rd ).walking time was increase with 10 min at 4 day and at 5th day stair climbing the ABGS was record in ICU 3 days.
  Interventions: Other: Continuous Positive Air Way Group
- Control Group (Active Comparator): Day 1: Bed mobility chest physiotherapy, active assistive ROM 5 repetitions of upper and lower limb, ACBT cycle. ABGS was analyses at first minute of exercise and vital was record after exercise.
  Day 2: Active range of motion exercise progress with 5 repetitions bed to chair mobility. same exercise progress with 5 repetition and 5 minute walk( day 3rd ).walking time will increase with 10 min at 4 day and at 5th day stair climbing the ABGS was record in ICU 3 days.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Continuous Positive Air Way Group — CPAP between 10 and 12 cmH2O
  Arms: Continuous Positive Air Way Group
Other: Control Group — Day 1: Bed mobility chest physiotherapy, active assistive ROM 5 repetitions of upper and lower limb, ACBT cycle. ABGS was analyses at first minute of exercise and vital was record after exercise.
  Day 2: Active range of motion exercise progress with 5 repetitions bed to chair mobility. same exercise progress with 5 repetition and 5 minute walk( day 3rd ).walking time will increase with 10 min at 4 day and at 5th day stair climbing the ABGS was record in ICU 3 days.
  Arms: Control Group

SUMMARY:
Different studies reported that CPAP is effective to prevent respiratory complication in post CABG patient and have greater impact on walking time, ventilatory function and breathing pattern.

DETAILED DESCRIPTION:
The walking time (6 minute walk test), effect on arterial blood gasses and long term effects of CPAP on cardiac activity, the previous studies focus only on the acute effects of CPAP along with specific exercises but did not tell about the long term effects. based on these finding this study is design to assess the effectiveness of CPAP in Post-op CABG patients regarding there early mobilization, walking time, ABGs and Ejection Fraction as there prognostic parameters in both phase-1 cardiac rehabilitation within hospital as well as in long-term prognosis, is of great interest.

ELIGIBILITY:
Inclusion Criteria:

* age between 35 to 60 years.
* With a clinical diagnosis of coronary artery disease, underwent elective CABG (Acute)

Exclusion Criteria:

* Low ejection friction (15%)
* Patient those who have any arrhythmias
* Unstable angina
* Patient having pace maker and implantable cardioverter defibrillator
* COPD and asthmatic patient
* Patient having BMI more then 40

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — clinical diagnosis of coronary artery disease, underwent elective CABG (Acute)
Enrollment: 38 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Arterial Blood Gasses | 3 days
  measures oxygen and carbon dioxide levels in your blood. It also measures your body's acid-base (pH) level, which is normally balanced when you are healthy.

SECONDARY OUTCOMES:
6 minute walk test | 3 days
  gold standard test to measure exercise capacity and requires less physical space and allows for easier monitoring of vital parameters
Ejection Fraction | 4 week
  expressed as a percentage, of how much blood the left ventricle pumps out with each contraction.
Short Form 12 Questionnaire | 4 weeks
  measuring tool for mental and physical health components. It consists of 12 questions which cover the eight health domain with one or two question per domain

CONTACTS AND LOCATIONS:
Overall Officials: Sumaiyah Obaid, MS, Principal Investigator — Riphah International University
Locations (1):
- Northwest General Hospital and research center, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No